CLINICAL TRIAL: NCT04124328
Title: The MARSHALINE Study: Evaluation of Vein of Marshall Ethanol Infusion During Left Atrial Linear Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Evaluation of Vein of Marshall Ethanol Infusion During Left Atrial Linear Ablation in Patients With Persistent Atrial Fibrillation
Acronym: MARSHALINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Professor Doctor, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2515
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALINE only group (Active Comparator): Patients in this arm are scheduled for an extended AF ablation, including the mitral isthmus line, according to the ALINE criteria
  Interventions: Procedure: ALINE only
- VoM group (Active Comparator): Patients in this arm are scheduled for an extended AF ablation, including the mitral isthmus line, according to the ALINE criteria and vein of Marshall (VoM) ethanol infusion
  Interventions: Procedure: ALINE + VoM infusion

INTERVENTIONS:
Procedure: ALINE + VoM infusion — In patients assigned to the ALINE + VoM infusion group, extended ablation will be performed according to the ALINE criteria. Additionally, the vein of Marshall will be infused with ethanol.
  Arms: VoM group
Procedure: ALINE only — In patients assigned to the ALINE only, extended ablation will be performed according to the ALINE criteria.
  Arms: ALINE only group

SUMMARY:
In this prospective, randomized, controlled, unblinded, mono-center study, we aim to evaluate the efficacy of vein of Marshall ethanol infusion during left atrial linear ablation in patients with atrial fibrillation compared to the ALINE protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 85 years
* Diagnosed with symptomatic AF without previous mitral isthmus line ablation

Exclusion Criteria:

* Previous MI line ablation
* Left atrial thrombus. LAA thrombus can be determined by preprocedural imaging: CT, TEE or MRI.
* LA diameter greater than 55 mm on long axis parasternal view, or left atrial volume more than 200 cc.
* Left ventricular ejection fraction <35%.
* Cardiac surgery within the previous 90 days.
* Expecting cardiac transplantation or other cardiac surgery within 180 days.
* Coronary PTCA/stenting within the previous 90 days or myocardial infarction within the previous 60 days.
* Documented history of a thromboembolic event within the previous 90 days.
* Diagnosed atrial myxoma.
* Significant restrictive, constrictive, or chronic obstructive pulmonary disease with chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Women who are pregnant or who plan to become pregnant during the study.
* Acute illness or active infection at time of index procedure
* Renal insufficiency
* Unstable angina.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation.
* Life expectancy less than 1 year.
* Uncontrolled heart failure.
* Presence of a condition that precludes vascular access.
* INR greater than 3.5 within 24 hours of procedure - for patients taking warfarin.
* Patient cannot be removed from antiarrhythmic drugs for reasons other than AF.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Procedural succes rate | At time of ablation
  Mitral isthmus block rate after one pass of the mitral line

SECONDARY OUTCOMES:
Total procedure time | At time of ablation
Fluoroscopy time | At time of ablation
Total RF ablation time | At time of ablation
Total extent of ablated LA tissue | At time of ablation
Cardiovascular-related hospitalizations | From time of ablation to one month post procedure
Changes in quality of life (SF36) | From inclusion to one month post procedure
Incidence of atrial flutter | From time of ablation to one month post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

REFERENCES:
- [Derived] Gillis K, O'Neill L, Wielandts JY, Hilfiker G, Almorad A, Lycke M, El Haddad M, le Polain de Waroux JB, Tavernier R, Duytschaever M, Knecht S. Vein of Marshall Ethanol Infusion as First Step for Mitral Isthmus Linear Ablation. JACC Clin Electrophysiol. 2022 Mar;8(3):367-376. doi: 10.1016/j.jacep.2021.11.019. Epub 2022 Feb 23. PMID 35331432